CLINICAL TRIAL: NCT02793323
Title: Superficial Cervical Nerve Block Versus NSAIDs for the Relief of Shoulder Tip Pain After Laparoscopic Surgeries
Brief Title: Superficial Cervical Nerve Block vs NSAIDs for the Relief of Shoulder Pain After Laparoscopic Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Zoher Naja, Chairperson of Anesthesia and Pain Management Department, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MakassedGH
Record Dates: First submitted 2016-05-30; First posted 2016-06-08 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Relieve Shoulder Pain After Laparoscopic Surgeries
MeSH Terms: interventions — Anti-Inflammatory Agents, Non-Steroidal; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Superficial cervical block (Experimental): Patients will receive superficial cervical nerve block in which we inject 5 ml of local anaesthetic mixture. Each 17 ml of the mixture contain: 6 ml lidocaine 2%, 6 ml lidocaine 2% with adrenaline 5 µg/ml, and 5 ml bupivacaine 0.5. Patients will also receive 100 ml IV saline.
  Interventions: Other: Superficial cervical nerve block; Other: General anesthesia; Other: IV placebo
- NSAID (Placebo Comparator): Patients will receive 100 mg (100 ml) IV NSAIDs (Profenid) before induction of anesthesia. Superficial cervical nerve block containing 5 ml placebo will be performed.
  Interventions: Other: NSAID; Other: General anesthesia; Other: Placebo superficial cervical nerve block

INTERVENTIONS:
Other: Superficial cervical nerve block — A nerve stimulator is used to guide superficial cervical blockade to relieve shoulder pain.
  Arms: Superficial cervical block
Other: NSAID — 100 mg (100 ml) intravenous NSAIDs (Profenid)
  Arms: NSAID
Other: General anesthesia — General anesthesia is induced with 1 μg/kg fentanyl, 1.5-2 mg/kg propofol and 1-2 mg midazolam. Then, endotracheal intubation is facilitated by 0.15 mg/kg nimbex. Anesthesia is maintained by 1-1.5% sevoflurane, 0.5 μg/kg/h fentanyl, 0.05 mg/kg/h nimbex, 60% nitrous oxide and 40% oxygen
Other: IV placebo — 100 ml IV saline
  Arms: Superficial cervical block
Other: Placebo superficial cervical nerve block — Superficial cervical nerve block containing 5 ml saline
  Arms: NSAID

SUMMARY:
Shoulder pain is frequently mentioned in recent literature following laparoscopic operations. Several pain relief strategies have been proposed to decrease shoulder tip pain post laparoscopic surgeries. This study will be conducted to compare the Superficial cervical nerve block vs. NSAIDs in terms of shoulder tip pain relief after laparoscopic surgeries.

DETAILED DESCRIPTION:
The study will be conducted in the operating room and post anesthesia care unit (PACU) at Makassed General Hospital. This is a prospective double blind randomized clinical trial that will be conducted between June 2016 and June 2017 at Makassed General Hospital. Following the Institutional Review Board (IRB) approval, written informed consent will be obtained from patients. Patients will be randomly assigned using the sealed envelope technique into 2 groups. Group I will receive superficial cervical nerve block and intravenous saline. Group II will receive saline superficial cervical block and intravenous NSAID (Profenid).

All patients will receive general anesthesia. General anesthesia is induced with 1 μg/kg fentanyl, 1.5-2 mg/kg propofol and 1-2 mg midazolam. Then, endotracheal intubation is facilitated by 0.15 mg/kg nimbex. Anesthesia is maintained by 1-1.5% sevoflurane, 0.5 μg/kg/h fentanyl, 0.05 mg/kg/h nimbex, 60% nitrous oxide and 40% oxygen. Any hemodynamic change of 25% results in a gradual increase or decrease of the sevoflurane concentration.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic:

cholecystectomy, sleeve gastrectomy, mini bypass surgery, gastric plication

Exclusion Criteria:

* Patients with kidney disease (ACUTE OR CHRONIC)
* Patients with allergy to any medication used throughout the research
* Patients with gastroesophageal reflux disease (GERD), peptic ulcer or duodenal ulcer disease
* Patients with shoulder neck pain or complications pre-operatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06-01; Primary Completion 2017-08-31 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Pain scores assessed through the Visual Analogue Scale (VAS) | 48 hours postoperatively

SECONDARY OUTCOMES:
Number of patients receiving analgesics | 48 hours postoperatively
Length of hospital stay | An average of 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Zoher Naja, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon